CLINICAL TRIAL: NCT06259916
Title: Developing Predictive Models to Distinguish Alcohol Use, Cannabis Use and Co-use: An Exploration of Electroencephalography (EEG) Metrics and Traditional Intoxication Measures
Brief Title: Distinguishing Alcohol Intoxication, Cannabis Intoxication and Co-intoxication Using Electroencephalography (EEG)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5061
Record Dates: First submitted 2024-01-09; First posted 2024-02-14 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Cannabis Use; Alcohol Use, Unspecified
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol; nabiximols

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cannabis Group (Experimental): Participants in this group will self-administer their own flower cannabis product (that they purchased for use in the study from a legal-market dispensary) ad libitum inside their homes. Researchers will not handle the product or instruct participants on how much to use during the session.
  Interventions: Other: Cannabis
- Alcohol Group (Experimental): Participants in this group will be administered a dose of alcohol by researchers in our mobile lab. The dose is designed (based on participant sex and body weight) to bring blood alcohol concentration to .06 g/dL.
  Interventions: Other: Alcohol
- Alcohol + Cannabis Group (Experimental): Participants in this group will first self-administer their own flower cannabis product (that they purchased for use in the study from a legal-market dispensary) ad libitum inside their homes. Researchers will not handle the product or instruct participants on how much to use during the session. They will then return to the mobile lab which will be parked outside their residence and will be administered a dose of alcohol by researchers. The dose is designed (based on participant sex and body weight) to bring blood alcohol concentration to .06 g/dL.
  Interventions: Other: Alcohol; Other: Cannabis

INTERVENTIONS:
Other: Alcohol — Participants in this condition will receive the standard alcohol dose
  Arms: Alcohol + Cannabis Group; Alcohol Group
Other: Cannabis — Participants in this group will self-administer legal-market flower cannabis
  Arms: Alcohol + Cannabis Group; Cannabis Group

SUMMARY:
This is a randomized, parallel-group study designed to explore the differences between cannabis intoxication, alcohol intoxication and co-intoxication involving both alcohol and cannabis, utilizing electroencephalography (EEG) as well as more traditional intoxication measures such as breath alcohol concentration and balance metrics. If eligible for the study, participants will be randomized to complete one study session in our mobile laboratory, during which they will use either alcohol, cannabis (which will be self-administered, ad libitum) or both alcohol and cannabis.

ELIGIBILITY:
Inclusion Criteria:

* 21-50 years old
* Heavy drinkers (consuming more than 4 drinks/day or more than 14 drinks/week for men, or more than 3 drinks/day or more than 7 drinks/week for women)
* Regular users of legal-market flower cannabis (at least 2x/week in past 3 months)
* report simultaneously using alcohol and legal-market flower cannabis at least once per month in the past 3 months
* English speakers.

Exclusion Criteria:

* Daily tobacco users
* Diagnosed with or seeking treatment for alcohol use disorder (AUD) or other substance use disorder (SUD)
* Females cannot be pregnant, breastfeeding or trying to become pregnant
* Meet criteria for psychotic, bipolar or major depressive disorder with suicidal ideation, or history of these disorders, 5) Current use of psychotropic (except anti-depressants)
* Report illicit drug use in past 60-days or fail drug screen on the day of the study appointment
* Major medical condition contraindicating alcohol and/or cannabis consumption.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography (EEG) Objective Cognitive Function Measures--Amplitude (microvolts) | Immediately pre-substance use, 1-hour post-use, 2-hours post-use, 4-hours post-use
  The EEG amplitude (measured in microvolts) will be obtained while participants perform the speeded visual flanker task
Electroencephalography (EEG) Objective Cognitive Function Measures--Latency (milliseconds) | Immediately pre-substance use, 1-hour post-use, 2-hours post-use, 4-hours post-use
  The EEG latency (measured in milliseconds) will be obtained while participants perform the speeded visual flanker task
Standing postural stability | Immediately pre-substance use, 1-hour post-use, 2-hours post-use, 4-hours post-use
  An iPod Touch will be attached to each participant's hip with a simple elastic/Velcro strap. An app on the device will record fine grained movements while they try to stand as still as possible for 30-60 seconds under four conditions that vary in terms of demand on the proprioceptive system (eyes open, eyes closed), and on a stable vs. soft (foam) surface.

OTHER OUTCOMES:
Breath Alcohol Concentration | Immediately pre-substance use, 1-hour post-use, 2-hours post-use, 4-hours post-use
  Measured using hand-held breathalyzer device
Blood Delta-9-tetrahydrocannabinol (THC) Levels | Immediately pre-substance use, 1-hour post-use, 2-hours post-use, 4-hours post-use
  THC measured from blood samples
Blood Cannabidiol (CBD) Levels | Immediately pre-substance use, 1-hour post-use, 2-hours post-use, 4-hours post-use
  CBD measured from blood samples
Blood Levels of 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol (THC-COOH) | Immediately pre-substance use, 1-hour post-use, 2-hours post-use, 4-hours post-use
  THC-COOH measured from blood samples
Blood Levels of 11-Hydroxy-Δ9-tetrahydrocannabinol (11-OH-THC) | Immediately pre-substance use, 1-hour post-use, 2-hours post-use, 4-hours post-use
  11-OH-THC measured from blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Hollis Karoly, PhD, Principal Investigator — Colorado State University; Patricia Davies, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States